CLINICAL TRIAL: NCT02946151
Title: Subcutaneous EEG in Epilepsy - Proof of Concept and Clinical Applications
Brief Title: Subcutaneous EEG in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: UNEEG Medical A/S (Industry); Technical University of Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016IL01; CIV-16-05-015704 (Other: EUDAMED)
Record Dates: First submitted 2016-10-19; First posted 2016-10-27 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Epilepsy; Seizure monitoring; Electroencephalography
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation (Experimental): Implantation of a subcutaneous electrode and connection to the external logging device
  Interventions: Device: UNEEG implantable EEG electrode and data storage device

INTERVENTIONS:
Device: UNEEG implantable EEG electrode and data storage device — The implantable EEG electrode will be implanted subcutaneously in the relevant temporal region by a certified neurosurgeon. The EEGgraphical data recorded will be transmitted transcutaneously to the data storage device via an inductive link, providing continuous data on brain activity.

SUMMARY:
The study is a two-phase study, which aims to explore the uses of a novel electrode type in detecting epileptic seizures. The electrode is designed for subcutaneous implantation with long-term monitoring in mind.

DETAILED DESCRIPTION:
The problem of unrecognized seizures is common for certain types of epilepsy. Electroencephalography (EEG) is an excellent method for seizure identification and recognition, but until now, it has not been feasible to perform EEG recordings for more than a few days outside a hospital or laboratory. A novel device has been developed, which might remedy that. The device is a EEG-electrode for subcutaneous implantation connected to an external data storage device.

The investigators in this study hypothesize that this device might be a useful tool for ultra-long-term epilepsy monitoring. The study aims to investigate that. While the device might be used to diagnose epilepsy, it is more likely to be a good seizure counting tool and that is what the study aims to determine.

Subjects include patients with mesial temporal lobe epilepsy and high seizure frequency. These will have the device implanted. Study phase 1 is a proof of concept to determine whether the device is actually able to detect epileptic seizures. This will take place during admission and be performed as simultaneous recordings with ordinary scalp EEG and the investigational device. Study phase 2 is a home monitoring to prove that devices actually provides clinically useful information regarding seizures in an outpatient setting.

The study requires 9 visits from each subject over the course of 4-6 months. The investigational device will be explanted after approximately 75 days of wear.

ELIGIBILITY:
Inclusion Criteria:

1. Semiology of some seizures compatible with mesial temporal lobe involvement.
2. Paraclinical findings supporting mesial temporal seizure focus. Such proof may consist of:

   * previous EEG recording interpreted as compatible with mesial temporal involvement OR
   * radiological findings demonstrating pathology in the mesial temporal area (CT, MRI, FDG-PET or SPECT).
3. Age 18-90.
4. Current seizure frequency (fulfilling criteria 1) of more than one per week to be eligible to EMU admission or 1 per month for direct enrollment to home monitoring (by own account).
5. Available for the duration of the study (6 months from screening).

Exclusion Criteria:

1. Known disorder of hemostasis.
2. Daily or frequent (more than 2 days per week) treatment with any drugs of the following types:

   * antiplatelets
   * anticoagulants
   * chemotherapeutics
   * non-steroid anti-inflammatory drugs (NSAID)
   * omega 3 fatty acids (fish oil)
3. Skeletal deformities or damage at the proposed implantation site to an extent that impedes correct electrode placement.
4. Scheduled facial or cranial surgery within 6 months from enrollment.
5. Active deep brain stimulation device.
6. Presence of implanted ICD pacemaker, cochlear implant or other active implants.
7. Planned transcranial magnetic stimulation (TMS) or transcranial direct current stimulation (tDCS) in the duration of the study.
8. Presence of any implanted device at the proposed site of implantation.
9. Known allergy towards any material that is part of the investigational device.
10. Females of childbearing potential who are pregnant, intend to become pregnant, or are not using adequate contraceptive methods throughout the study.
11. Performing extreme sport, including scuba diving (snorkel diving is allowed), parachute jumping or martial arts.
12. Scheduled MRI within 5 months from enrollment.
13. Work involving operation of MRI-scanner.
14. Operating hand held transceivers for communication (e.g. within the police, medical, fire, air traffic control, marine or military).
15. Working at broadcast stations for television or FM/DAB radio.
16. Known or suspected abuse of alcohol defined as estimated consumption beyond that, which is recommended by the DHA or any other neuro-active substances.
17. Active vagus nerve stimulator.
18. Skin disorders near the proposed implantation site, including infection.
19. Contraindications against the local anesthetic drug used during im- and explantation.
20. Diabetes of any kind.
21. Psychiatric disorders including:

    * schizophrenia
    * bipolar affective disorder
    * emotionally unstable personality disorder
    * schizoaffective disorder
    * schizotypal disorder
    * autism
22. Severely abnormal paraclinical findings or vital signs:

    * S-creatinine ≥ 3 times upper reference value
    * ALAT, alkaline phosphatase or bilirubin≥ 3 times upper reference value
    * APTT > 50 seconds
    * thrombocyte count < 50 or >1000 x 10^9/l
    * INR ≥ 1,6
    * HgBA1C > 55 mmol/mol
    * Any ECG finding requiring immediate referral to a cardiologist as assessed by the investigator
    * pulse <40 bpm or >120 bpm or suspicion of atrial fibrillation by auscultation
    * temperature >38 ºC
    * respiration rate >30 pr. minute
    * systolic blood pressure < 80 mmHg or >220 mmHg and diastolic blood pressure <50 mmHg or >120 mmHg
    * any other clinical or paraclinical finding suggesting known or unknown illness or disorder requiring immediate treatment as assessed by the investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11; Primary Completion 2019-01-23 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Seizure comparison | 24 months
  Qualitative comparison of patient-recorded seizures and EEGgraphical seizures
Adverse events | 24 months
  Descriptive account of device related adverse events
Compliance | 24 months
  Descriptive account of compliance in use of the investigational device

CONTACTS AND LOCATIONS:
Overall Officials: Troels Kjær, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gangstad SW, Mikkelsen KB, Kidmose P, Tabar YR, Weisdorf S, Lauritzen MH, Hemmsen MC, Hansen LK, Kjaer TW, Duun-Henriksen J. Automatic sleep stage classification based on subcutaneous EEG in patients with epilepsy. Biomed Eng Online. 2019 Oct 30;18(1):106. doi: 10.1186/s12938-019-0725-3. PMID 31666082